CLINICAL TRIAL: NCT04843683
Title: StereoTactic Ablative RadioTherapy of Cardiac Arrhythmias (START-CA): a Phase II Trial of Non-Invasive Treatment of Medically Refractory Patients
Brief Title: StereoTactic Ablative RadioTherapy of Cardiac Arrhythmias (START-CA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-6027
Record Dates: First submitted 2021-04-01; First posted 2021-04-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic ablative radiotherapy (SBRT) Arm (Experimental): Stereotactic ablative radiotherapy (SBRT) is a type of radiation treatment that delivers precise, high dose radiation to targeted areas. In this study, a single treatment of SBRT will be delivered to the abnormal area of a participant's heart that is causing dangerous heart rate and rhythm changes (arrhythmia).
  Interventions: Radiation: Stereotactic Ablative Radiotherapy
- Observational Arm (No Intervention): Potential participants who are eligible to be included in the study, but who choose not to have the SBRT procedure, can still receive standard medical treatment alone and be followed up with study visits and questionnaires.

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy — Stereotactic ablative radiotherapy (SBRT) is a type of radiation treatment that delivers precise, high dose radiation to targeted areas. In this study, a single treatment of SBRT will be delivered to the abnormal area of a participant's heart that is causing dangerous heart rate and rhythm changes (arrhythmia).
  Arms: Stereotactic ablative radiotherapy (SBRT) Arm

SUMMARY:
This is a prospective, single-center, phase II trial that will be monitoring the safety and efficacy of using stereotactic ablative radiotherapy (SBRT) to treat patients with a medical condition affecting heart rate and rhythm (refractory arrhythmias) within the University Health Network (Princess Margaret Cancer Centre and Toronto General Hospital). The primary objective will be to prospectively monitor patient cardiac outcomes following SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart rate and rhythm condition (arrhythmia) who have failed standard of care treatment with medication OR at least one prior invasive catheter ablation procedure.
* Patients deemed medically fit to receive stereotactic ablative radiotherapy as determined by their Radiation Oncologist.

Exclusion Criteria:

* Patients who have previously received high dose radiotherapy to the target area and cannot safely receive further treatment OR are unable to receive radiotherapy due to other contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in ICD therapies. | Baseline to 18 months follow-up.
  Patient cardiac outcomes will be evaluated by changes from baseline in ICD (Implantable Cardioverter-Defibrillator) therapies (ICD shock frequency) following radiotherapy at 1, 3, 6, 12 and 18 months of follow-up.
Change from Baseline in the number or dose of antiarrhythmic medications. | Baseline to 18 months follow-up.
  Patient cardiac outcomes will be evaluated by changes from baseline in the number or dose of antiarrhythmic medications following radiotherapy at 1, 3, 6, 12 and 18 months of follow-up.

SECONDARY OUTCOMES:
Measure patient quality-of-life during the study. | Baseline to 18 months follow-up.
  Patient-Reported Health Related Quality of Life (HRQOL) will be assessed at each 1, 3, 6, 12 and 18 month follow-up, using the following assessment questionnaires: 36-item Short Form Health Survey (SF-36).
Measure patient quality-of-life during the study. | Baseline to 18 months follow-up.
  Patient-Reported Health Related Quality of Life (HRQOL) will be assessed at each 1, 3, 6, 12 and 18 month follow-up, using the following assessment questionnaire: the Hospital Anxiety and Depression Scale (HADS-A). A lower score indicates a better outcome.
  HADS-A Scoring: 0-7 = Normal, 8-10 = Borderline abnormal (borderline case), 11-21 = Abnormal (case).
Measure patient subjective distress following treatment. | Baseline to 6 months follow-up
  Patient subjective distress following treatment will be measured at baseline, and 1 month and 6-months follow-up, using the Impact of Events Scale (IES-R). A higher score indicates a worse outcome.
  IES-R Scoring: 24 or more = Post-traumatic stress disorder (PTSD) is a clinical concern. 33 and above = This represents the best cutoff for a probable diagnosis of PTSD. 37 or more = This is high enough to suppress immune system's functioning.
Overall mortality record. | 6 to 18 months follow-up.
  Safety will be evaluated by recording overall mortality at 6 month intervals post-treatment.
Number of patients with acute and long-term toxicity as assessed by CTCAE v5.0. | 1 month to 18 months follow-up.
  Acute (less than or equal to 90 days) and long-term (greater than 90 days) toxicity will be evaluated by using prospective follow-up and grading according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Rates of hospital admissions. | Baseline to 18 months follow-up.
  Safety will be evaluated by recording rates of hospital admission during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Center, University Health Network, Toronto, Ontario, Canada